CLINICAL TRIAL: NCT00522769
Title: Development of CBT Model for Adolescent Bulimia Nervosa
Brief Title: Cognitive Behavioral Therapy to Treat Bulimia Nervosa in Adolescents
Acronym: claire
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Lynn DeBar, PhD MPH, Kaiser Permanente
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5R34MH073796 (NIH)
Record Dates: First submitted 2007-08-29; First posted 2007-08-30 (Estimated); Last update posted 2010-02-15 (Estimated); Status verified 2010-02

CONDITIONS: Bulimia Nervosa
Keywords: binge eating; adolescent girls; cognitive behavioral therapy
MeSH Terms: conditions — Bulimia Nervosa; Bulimia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Delayed Intervention (Active Comparator): 1/2 of participants are randomized to immediate intervention that starts within a week of randomization. The other 1/2 of the participants are randomized to delayed intervention which starts 6 months after randomization.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Immediate intervention (Experimental): Immediate intervention starts within two weeks of randomization. Delayed interventions starts 6 months after randomization.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Girls enrolled in the study will either receive the 6-20 session CBT intervention at the time of enrollment or 6 months after they enroll. Assessments including questions about eating behaviors, mood, and general functioning are given on enrollment in the study, and 3- and 6-months following enrollment (also at 9- and 12-months for those in the delayed treatment condition

SUMMARY:
The claire project is a research study testing the use of Cognitive Behavioral Therapy (CBT) to help teenage girls develop healthier eating habits and better ways to manage weight and shape concerns. The study is enrolling girls who are members of the Kaiser Permanente Health plan in the Northwest region. They must be between the ages of 12 and 18 and report binge eating and/or purging (vomiting, laxative or diuretic use) at a research established threshold to be eligible for the study. Girls enrolled in the study will either receive the 6-20 session CBT intervention at the time of enrollment or 6 months after they enroll. Assessments including questions about eating behaviors, mood, and general functioning are given on enrollment in the study, and 3- and 6-months following enrollment (also at 9- and 12-months for those in the delayed treatment condition).

DETAILED DESCRIPTION:
The overall aim of this study is to develop a manual-based cognitive behavioral therapy (CBT) intervention to treat bulimia nervosa spectrum conditions (BN and EDNOS) in adolescents identified with these conditions in a large HMO in the Pacific Northwest. Eating disorders are among the most common, impairing, and serious mental health problems-particularly among women. BN and its subclinical variants usually arise in adolescence and affects as many as 10% of young women. Yet despite the significance of these conditions, there are no systematic studies of empirically-based interventions for adolescents with BN and EDNOS. We propose to design an intervention based on the adult CBT model, addressing developmental considerations of adolescents, as well as the risk and maintaining factors of adolescent BN/EDNOS. In addition to developing the adolescent-specific CBT protocol, we will evaluate adolescent, family, and medical provider satisfaction with this intervention. We will estimate effect-size and effect-size variability of this intervention's impact on primary (binge and purge cessation and frequency) and secondary outcomes measured post-treatment and at a 6-month follow-up. These results will inform a subsequent, full-scale, randomized clinical trial. We will develop the intervention in two distinct phases. The first phase (months 1 to 18) will consist of at least two development cycles of the adolescent BN-CBT program. In each cycle, we will draft a version of the intervention, test it with several clinical cases, obtain feedback from adolescents and their parents, and then generate a new version of the intervention. We will start with a 6-20 session adaptation of the Fairburn, Marcus, and Wilson (1993) CBT intervention, and modify it to fit an adolescent population. The development and revision process will be led by our core Expert Group of clinicians and researchers meeting weekly. We will be guided by the Expert Group's prior experiences developing and evaluating CBT for adult BN, and CBT for adolescent depression; and qualitative feedback from youth, parent, and provider stakeholders. In the second phase (months 19 to 32), we will conduct a larger pilot for the purpose of estimating effect size, using the stable, final version of the intervention. The pilot will enroll 50 adolescents and their families who are identified through their pediatric providers in the HMO or in response to a mass mailing of recruitment materials and a screening questionnaire. Half of the participants will be randomized to receive the intervention immediately upon enrollment and half (Wait List) to a treatment as usual followed by a delayed intervention 6 months after enrollment. Data will be collected through interviews with the teen and a parent at baseline, 3 months, 6 months and for the Wait List teens, at 9 months and 12 months post enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 12-18, inclusive.
2. Female
3. A DSM-IV diagnosis of current BN or spectrum BN
4. One or both parent(s) willing to participate in study assessments and intervention visit

Exclusion Criteria:

1. A current DSM-IV diagnosis of AN.
2. A DSM-IV diagnosis of a psychotic disorder (current or past).
3. Current or past cognitive behavior therapy for an eating disorder or other mental health condition
4. Currently receiving antidepressant medication or medications known to impact weight
5. A significant organic brain syndrome, mental retardation, pervasive developmental disorder or autism.
6. Current pregnancy.
7. Current treatment specifically for ED (not counting medical case management).

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2005-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Recovery from ED (abstinence of all binging and purging during past 28 indices of binge eating, purging, and scores on the EDE-Q5 scale). | 6 months

SECONDARY OUTCOMES:
: changes in other psychiatric symptomatology and | 6 months
associated adaptive functioning and eating concerns | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lynn L DeBar, PhD MPH, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente Center for Health Research, Portland, Oregon, United States